CLINICAL TRIAL: NCT03295513
Title: Clinical Evaluation of Wear Behavior of Human Enamel and Chipping of Veneered Zirconia Against Monolithic Zirconia (Randomized Controlled Clinical Trial)
Brief Title: Clinical Evaluation of Wear Behavior of Human Enamel and Chipping of Veneered Zirconia Against Monolithic Zirconia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nouran Mahmoud Ibrahim Metwally, mSc, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CEBD-CU-2017-09-21
Record Dates: First submitted 2017-09-15; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Broken Tooth With Complication; Non Vital Teeth; Mutilated Teeth
Keywords: mutilated, root canal treated teeth, and coronal fracture

STUDY DESIGN:
Intervention Model Description: Patient will receive a restoration with superior function, esthetics, and quality.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- veneered zirconia full coverage restorations (Active Comparator): InCoris zirconia material (TZI-Densupply sirona)
  Interventions: Other: Veneered zirconia
- Monolithic zirconia full coverage restorations (Experimental): InCoris (TZI-Densupply sirona)
  Interventions: Other: Monolithic zirconia

INTERVENTIONS:
Other: Veneered zirconia — he use of veneered zirconia is well documented in the literatures as successful restoration modality. A two Clinical performance of two different CAD/CAM-fabricated ceramic crowns revealed no chipping for veneered zirconia
  Arms: veneered zirconia full coverage restorations
Other: Monolithic zirconia — Monolithic zirconia product presented a new generation of polycrystalline material by which full anatomical crowns and bridges can be produced
  Arms: Monolithic zirconia full coverage restorations

SUMMARY:
The aim of this study is to evaluate chipping and the degree of natural enamel loss opposing to monolithic zirconia compared to veneered zirconia restoration.

DETAILED DESCRIPTION:
While increase using of zirconia in extra coronal restoration as a substitute for metal ceramic restoration still high rate of technical complications specifically chipping of veneering ceramic and wear of antagonist are usually associated with veneered zirconia restoration which led to development of new monolithic zirconia to overcome these technical complications.

Therefore this study will be conducted to evaluate chipping and wear of antagonist of veneered zirconia versus monolithic zirconia all ceramic crowns in posterior area.

Benefits of the research to the patient:

Patient will receive a restoration with superior function, esthetics, and quality.

It will save teeth such as mutilated teeth, endodontically treated and teeth with massive loss of tooth structure that cannot be restored with direct restoration.

As a result of properly functioning restoration, teeth will be restored with predictable prognosis and the patient will be psychologically improved.

Benefits of the research to the clinician:

Practitioner will have the advantage to clinically assess a new material that can be used in different situations for better function and esthetic outcomes.

It will improve patient confidence with the dentist.

Explanation for choice of comparators:

The use of veneered zirconia is well documented in the literatures as successful restoration modality. A two Clinical performance of two different CAD/CAM-fabricated ceramic crowns revealed no chipping for veneered zirconia.

A 3 years Randomized Controlled Clinical Trial of Zirconia-Ceramic and Metal-Ceramic Posterior Fixed Dental Prostheses reported Alpha Scores A=66.6%, B =25% , C=5.6% and Only D= 2.8 A 5 years prospective clinical study of posterior zirconia fixed dental prosthesis reported Alpha scores greater than 95% indicating no predictable changes during the 5 years Another 3 years Randomized controlled clinical Trial of Posterior veneered zirconia for fixed dental prostheses revealed 20% chipping and also 30% reported alpha for antagonist wear and 70% reported bravo after 3 years of clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of the patients from 20-60 years old; able to read and sign the informed consent document, illiterate patient will be avoided.
2. Patients able physically and psychologically to tolerate conventional restorative procedures.
3. Patients with no active periodontal or pulpal diseases, having teeth with good restorations.
4. Patients with teeth problems indicated for full coverage restoration (e.g. Moderate to severe discoloration, coronal fracture where partial coverage would lack retention, malposed or malformed teeth).
5. Patients with root canal treated teeth requiring full coverage restorations.
6. Patients willing to return for follow-up examinations and evaluation.

Exclusion Criteria:

1. Patients in the growth stage with partially erupted teeth.
2. Patients with poor oral hygiene and motivation.
3. A pregnant woman's to avoid any complication that may occur in dental office due to pregnancy or due to injected anesthetic solution.
4. Patients with psychiatric problems or unrealistic expectation (patient that has phobia from dental treatments or needle bunch).
5. Patients have no opposite occluding dentition in the area intended for restoration.
6. Patients suffer from Para functional habits.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Chipping | 12 month
  chipping of the restoration by modified USPHs criteria as Alpha (Excellent) ideal,Bravo (Acceptable) less than ideal but no modifications required, Charlie (Acceptable but modifications needed) staining or other shade modifications required, and Delta (Unacceptable) remake.

SECONDARY OUTCOMES:
tooth wear | 12 month
  Measuring the effect on natural tooth by modified USPHs criteria as Alpha(Excellent) ideal,Bravo (Acceptable) less than ideal but no modifications requiredCharlie (Acceptable but modifications needed) staining or other shade modifications required, and Delta (Unacceptable) remake.